CLINICAL TRIAL: NCT04611399
Title: MIND-VR: Virtual Reality for COVID-19 Operators' Psychological Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIND-VR/Besta
Record Dates: First submitted 2020-10-08; First posted 2020-11-02 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-01

CONDITIONS: Stress Related Disorder
Keywords: virtual reality; stress; anxiety; prevention; treatment; relaxation techniques; psychoeducation; COVID-19; healthcare workers
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: The study can be defined as a controlled and randomized clinical trial, single-blind and monocentric, aimed at studying the efficacy of the intervention with virtual reality contents in reducing stress and anxiety in healthcare personnel involved in the care of COVID-19 patients. The study will be conducted according to the indications of Good Clinical Practices. The clinical efficacy of the intervention will be assessed at two different time distances (T0, T1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) Group (Experimental): The treatment for the participants allocated to the VR Group consists of three home-sessions of approximately 30 minutes each, conducted over one week. In each session, participants will be asked to try for about 15 minutes "MIND-VR". Subsequently, they will try the virtual relaxation content "The Secret Garden".
  Interventions: Behavioral: VR for psychoeducation and relaxation
- Control (CR) Group (Active Comparator): The CR Group will undergo pre- and post-protocol tests without undergoing any treatment.
  Interventions: Other: Control (CR)

INTERVENTIONS:
Behavioral: VR for psychoeducation and relaxation — Use of specifically developed VR contents to deliver psychoeducational content on stress and anxiety (i.e., "MIND-VR") and to train on relaxation techniques (i.e., "The Secret Garden").
  Arms: Virtual Reality (VR) Group
Other: Control (CR) — The CR Group will undergo pre- and post-protocol tests without undergoing any treatment.
  Arms: Control (CR) Group

SUMMARY:
Since the COVID-19 pandemic began, several psychological support programs for health care workers have been implemented, especially group or individual counseling sessions delivered face-to-face or using phones and video conferencing platforms. However, there are significant barriers to the delivery of such psychological initiatives. In this context, digital interventions to improve health services and care outcomes are recommended for implementing and providing remote psychological support. Virtual reality can play a relevant role in providing psychological care to healthcare workers facing COVID-19. New commercial head-mounted display have made virtual reality accessible even to the mass audience, breaking down the barriers in the diffusion and use of this technology. Thanks to this fact, virtual reality can now be autonomously used by people and offered to provide psychological assistance remotely. Within this context, this randomized controlled study aims to investigate the efficacy of a virtual reality home-based program for diminishing stress and anxiety in a sample of Italian healthcare workers involved in the COVID-19 pandemic.

DETAILED DESCRIPTION:
Since the COVID-19 pandemic began, several psychological support programs for health care workers have been implemented, especially group or individual counseling sessions delivered face-to-face or using phones and video conferencing platforms. However, there are significant barriers to the delivery of such psychological initiatives. In this context, digital interventions to improve health services and care outcomes are recommended for implementing and providing remote psychological support.

Virtual reality can play a relevant role in providing psychological care to healthcare workers facing COVID-19. New commercial head-mounted display have made virtual reality accessible even to the mass audience, breaking down the barriers in the diffusion and use of this technology. Thanks to this fact, virtual reality can now be autonomously used by people and offered to provide psychological assistance remotely.

Within this context, this randomized controlled trial (RCT) aims to investigate the efficacy of a virtual reality home-based program for diminishing stress and anxiety in a sample of Italian healthcare workers involved in the COVID-19 pandemic. In particular, the objective is to compare the efficacy of this type of training with respect to the same program without virtual reality and a waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, < 65;
* Having worked on the front line as a doctor or nurse during the COVID-19 emergency (i.e., having assisted COVID-19 patients or having worked in departments dedicated to COVID-19 patients);
* Normal or corrected to normal visual acuity;
* Normal or corrected to normal hearing ability.

Exclusion Criteria:

* Physical illness: cardiovascular issues, neurological illness, epilepsy;
* Pharmacotherapy with: psychotropic drugs, anti-hypertensive drugs, anti-epileptics;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Change in score at the State-Trait Anxiety Inventory -Y2 | Baseline; immediately after the procedure/intervention; 3 months and 6 months follow-up
  A 20 item measure of the level of the state anxiety
Change in score at the Perceived Stress Scale | Baseline; immediately after the procedure/intervention; 3 months and 6 months follow-up
  A 10 item measure of the level of stress perceived in the last month
Change in score at the Depression, Anxiety ans Stress Scale-21 items | Baseline; immediately after the procedure/intervention; 3 months and 6 months follow-up
  A 21 item in 3 self-report scales which measures depression, anxiety and stress
Change in score of knowledge on stress and anxiety | Baseline; immediately after the procedure/intervention; 3 months and 6 months follow-up
  A 7 item measure at the ad hoc questionnaire to assess the knowledge of stress and anxiety

SECONDARY OUTCOMES:
Change in score at the EQ-5D-5L | Baseline; immediately after the procedure/intervention; 3 months and 6 months follow-up
  A measure which defines the state of health and the perceived quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Federica Pallavicini, PhD, Study Director — University of Milano Bicocca; Eleonora F Orena, PhD, Principal Investigator — Foundation IRCCS Neurological Institute Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

REFERENCES:
- [Background] Anderson AP, Mayer MD, Fellows AM, Cowan DR, Hegel MT, Buckey JC. Relaxation with Immersive Natural Scenes Presented Using Virtual Reality. Aerosp Med Hum Perform. 2017 Jun 1;88(6):520-526. doi: 10.3357/AMHP.4747.2017. PMID 28539139
- [Background] Anderson E, Shivakumar G. Effects of exercise and physical activity on anxiety. Front Psychiatry. 2013 Apr 23;4:27. doi: 10.3389/fpsyt.2013.00027. eCollection 2013. No abstract available. PMID 23630504
- [Background] Bailenson, J. N., Yee, N., Blascovich, J., Beall, A. C., Lundblad, N., & Jin, M. (2008). The Use of Immersive Virtual Reality in the Learning Sciences: Digital Transformations of Teachers, Students, and Social Context. Journal of the Learning Sciences, 17(1), 102-141.
- [Background] Bakker M, Wicherts JM. The (mis)reporting of statistical results in psychology journals. Behav Res Methods. 2011 Sep;43(3):666-78. doi: 10.3758/s13428-011-0089-5. PMID 21494917
- [Background] Bangor, A., Kortum, P. T., & Miller, J. T. (2008). An Empirical Evaluation of the System Usability Scale. International Journal of Human-Computer Interaction, 24(6), 574-594.
- [Background] Basso JC, Suzuki WA. The Effects of Acute Exercise on Mood, Cognition, Neurophysiology, and Neurochemical Pathways: A Review. Brain Plast. 2017 Mar 28;2(2):127-152. doi: 10.3233/BPL-160040. PMID 29765853
- [Background] Beck JG, Palyo SA, Winer EH, Schwagler BE, Ang EJ. Virtual Reality Exposure Therapy for PTSD symptoms after a road accident: an uncontrolled case series. Behav Ther. 2007 Mar;38(1):39-48. doi: 10.1016/j.beth.2006.04.001. Epub 2006 Sep 22. PMID 17292693
- [Background] Botella C, Serrano B, Banos RM, Garcia-Palacios A. Virtual reality exposure-based therapy for the treatment of post-traumatic stress disorder: a review of its efficacy, the adequacy of the treatment protocol, and its acceptability. Neuropsychiatr Dis Treat. 2015 Oct 3;11:2533-45. doi: 10.2147/NDT.S89542. eCollection 2015. PMID 26491332
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] Chen Q, Liang M, Li Y, Guo J, Fei D, Wang L, He L, Sheng C, Cai Y, Li X, Wang J, Zhang Z. Mental health care for medical staff in China during the COVID-19 outbreak. Lancet Psychiatry. 2020 Apr;7(4):e15-e16. doi: 10.1016/S2215-0366(20)30078-X. Epub 2020 Feb 19. No abstract available. PMID 32085839
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] De Freitas, S., Rebolledo-Mendez, G., Liarokapis, F., Magoulas, G., & Poulovassilis, A. (2010). Learning as immersive experiences: Using the four-dimensional framework for designing and evaluating immersive learning experiences in a virtual world. British Journal of Educational Technology, 41(1),69-85.
- [Background] Difede J, Cukor J, Jayasinghe N, Patt I, Jedel S, Spielman L, Giosan C, Hoffman HG. Virtual reality exposure therapy for the treatment of posttraumatic stress disorder following September 11, 2001. J Clin Psychiatry. 2007 Nov;68(11):1639-47. PMID 18052556
- [Background] Difede J, Cukor J, Wyka K, Olden M, Hoffman H, Lee FS, Altemus M. D-cycloserine augmentation of exposure therapy for post-traumatic stress disorder: a pilot randomized clinical trial. Neuropsychopharmacology. 2014 Apr;39(5):1052-8. doi: 10.1038/npp.2013.317. Epub 2013 Nov 12. PMID 24217129
- [Background] Duan YY, Zhang JY, Xie M, Feng XB, Xu S, Ye ZW. Application of Virtual Reality Technology in Disaster Medicine. Curr Med Sci. 2019 Oct;39(5):690-694. doi: 10.1007/s11596-019-2093-4. Epub 2019 Oct 14. PMID 31612384
- [Background] Fish, M. T., Russoniello, C. V., & O'Brien, K. (2018). Zombies vs. Anxiety: An Augmentation Study of Prescribed Video Game Play Compared to Medication in Reducing Anxiety Symptoms. Simulation & Gaming, 49(5), 553-566.
- [Background] Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am Psychol. 2001 Mar;56(3):218-26. doi: 10.1037//0003-066x.56.3.218. PMID 11315248
- [Background] Fujii S, Kato H, Maeda K. A simple interview-format screening measure for disaster mental health: an instrument newly developed after the 1995 Great Hanshin Earthquake in Japan--the Screening Questionnaire for Disaster Mental Health (SQD). Kobe J Med Sci. 2008 Feb 8;53(6):375-85. PMID 18762732
- [Background] Gaggioli A, Pallavicini F, Morganti L, Serino S, Scaratti C, Briguglio M, Crifaci G, Vetrano N, Giulintano A, Bernava G, Tartarisco G, Pioggia G, Raspelli S, Cipresso P, Vigna C, Grassi A, Baruffi M, Wiederhold B, Riva G. Experiential virtual scenarios with real-time monitoring (interreality) for the management of psychological stress: a block randomized controlled trial. J Med Internet Res. 2014 Jul 8;16(7):e167. doi: 10.2196/jmir.3235. PMID 25004803
- [Background] Gerardi M, Rothbaum BO, Ressler K, Heekin M, Rizzo A. Virtual reality exposure therapy using a virtual Iraq: case report. J Trauma Stress. 2008 Apr;21(2):209-13. doi: 10.1002/jts.20331. PMID 18404648
- [Background] Gorini A, Griez E, Petrova A, Riva G. Assessment of the emotional responses produced by exposure to real food, virtual food and photographs of food in patients affected by eating disorders. Ann Gen Psychiatry. 2010 Jul 5;9:30. doi: 10.1186/1744-859X-9-30. PMID 20602749
- [Background] Gradl, S., Wirth, M., Zillig, T., & Eskofier, B. M. (2018). Visualization of heart activity in virtual reality: A biofeedback application using wearable sensors. In 2018 IEEE 15th International Conference on Wearable and Implantable Body Sensor Networks (BSN) (pp. 152-155). IEEE.
- [Background] Granic I, Lobel A, Engels RC. The benefits of playing video games. Am Psychol. 2014 Jan;69(1):66-78. doi: 10.1037/a0034857. Epub 2013 Dec 2. PMID 24295515
- [Background] Greenberg N, Docherty M, Gnanapragasam S, Wessely S. Managing mental health challenges faced by healthcare workers during covid-19 pandemic. BMJ. 2020 Mar 26;368:m1211. doi: 10.1136/bmj.m1211. No abstract available. PMID 32217624
- [Background] Heiman, G. W. (1998). Understanding research methods and statistics : an integrated introduction for psychology.
- [Background] Hoffman HG. Virtual-reality therapy. Sci Am. 2004 Aug;291(2):58-65. doi: 10.1038/scientificamerican0804-58. No abstract available. PMID 15298120
- [Background] Huang JZ, Han MF, Luo TD, Ren AK, Zhou XP. [Mental health survey of medical staff in a tertiary infectious disease hospital for COVID-19]. Zhonghua Lao Dong Wei Sheng Zhi Ye Bing Za Zhi. 2020 Mar 20;38(3):192-195. doi: 10.3760/cma.j.cn121094-20200219-00063. Chinese. PMID 32131151
- [Background] Kang L, Li Y, Hu S, Chen M, Yang C, Yang BX, Wang Y, Hu J, Lai J, Ma X, Chen J, Guan L, Wang G, Ma H, Liu Z. The mental health of medical workers in Wuhan, China dealing with the 2019 novel coronavirus. Lancet Psychiatry. 2020 Mar;7(3):e14. doi: 10.1016/S2215-0366(20)30047-X. Epub 2020 Feb 5. No abstract available. PMID 32035030
- [Background] Lee KM, Gilmore DF. Statistical experimental design for bioprocess modeling and optimization analysis: repeated-measures method for dynamic biotechnology process. Appl Biochem Biotechnol. 2006 Nov;135(2):101-16. doi: 10.1385/abab:135:2:101. PMID 17159235
- [Background] Li Z, Ge J, Yang M, Feng J, Qiao M, Jiang R, Bi J, Zhan G, Xu X, Wang L, Zhou Q, Zhou C, Pan Y, Liu S, Zhang H, Yang J, Zhu B, Hu Y, Hashimoto K, Jia Y, Wang H, Wang R, Liu C, Yang C. Vicarious traumatization in the general public, members, and non-members of medical teams aiding in COVID-19 control. Brain Behav Immun. 2020 Aug;88:916-919. doi: 10.1016/j.bbi.2020.03.007. Epub 2020 Mar 10. PMID 32169498
- [Background] Lindner P, Miloff A, Hamilton W, Carlbring P. The Potential of Consumer-Targeted Virtual Reality Relaxation Applications: Descriptive Usage, Uptake and Application Performance Statistics for a First-Generation Application. Front Psychol. 2019 Feb 4;10:132. doi: 10.3389/fpsyg.2019.00132. eCollection 2019. PMID 30778311
- [Background] Liu CY, Yang YZ, Zhang XM, Xu X, Dou QL, Zhang WW, Cheng ASK. The prevalence and influencing factors in anxiety in medical workers fighting COVID-19 in China: a cross-sectional survey. Epidemiol Infect. 2020 May 20;148:e98. doi: 10.1017/S0950268820001107. PMID 32430088
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Maples-Keller JL, Bunnell BE, Kim SJ, Rothbaum BO. The Use of Virtual Reality Technology in the Treatment of Anxiety and Other Psychiatric Disorders. Harv Rev Psychiatry. 2017 May/Jun;25(3):103-113. doi: 10.1097/HRP.0000000000000138. PMID 28475502
- [Background] McAlonan GM, Lee AM, Cheung V, Cheung C, Tsang KW, Sham PC, Chua SE, Wong JG. Immediate and sustained psychological impact of an emerging infectious disease outbreak on health care workers. Can J Psychiatry. 2007 Apr;52(4):241-7. doi: 10.1177/070674370705200406. PMID 17500305
- [Background] McLay RN, Wood DP, Webb-Murphy JA, Spira JL, Wiederhold MD, Pyne JM, Wiederhold BK. A randomized, controlled trial of virtual reality-graded exposure therapy for post-traumatic stress disorder in active duty service members with combat-related post-traumatic stress disorder. Cyberpsychol Behav Soc Netw. 2011 Apr;14(4):223-9. doi: 10.1089/cyber.2011.0003. Epub 2011 Feb 20. PMID 21332375
- [Background] Oing T, Prescott J. Implementations of Virtual Reality for Anxiety-Related Disorders: Systematic Review. JMIR Serious Games. 2018 Nov 7;6(4):e10965. doi: 10.2196/10965. PMID 30404770
- [Background] Pallavicini F, Gaggioli A, Raspelli S, Cipresso P, Serino S, Vigna C, Grassi A, Morganti L, Baruffi M, Wiederhold B, Riva G. Interreality for the management and training of psychological stress: study protocol for a randomized controlled trial. Trials. 2013 Jun 28;14:191. doi: 10.1186/1745-6215-14-191. PMID 23806013
- [Background] Pallavicini, F., Algeri, D., Repetto, C., Gorini, A., & Riva, G. (2009). Biofeedback, virtual reality and mobile phones in the treatment of generalized anxiety disorder (gad): A phase-2 controlled clinical trial. Journal of Cyber Therapy and Rehabilitation, 2(4), 315-327.
- [Background] Pallavicini F, Cipresso P, Raspelli S, Grassi A, Serino S, Vigna C, Triberti S, Villamira M, Gaggioli A, Riva G. Is virtual reality always an effective stressors for exposure treatments? Some insights from a controlled trial. BMC Psychiatry. 2013 Feb 11;13:52. doi: 10.1186/1471-244X-13-52. PMID 23398927
- [Background] Pallavicini, F., Ferrari, A., Zini, A., Garcea, G., Zanacchi, A., Barone, G., & Mantovani, F. (2018). What Distinguishes a Traditional Gaming Experience from One in Virtual Reality? An Exploratory Study (pp. 225-231). Springer, Cham.
- [Background] Pallavicini, F., & Pepe, A. (2019). Comparing Player Experience in Video Games Played in Virtual Reality or on Desktop Displays. In Extended Abstracts of the Annual Symposium on Computer-Human Interaction in Play Companion Extended Abstracts - CHI PLAY '19 Extended Abstracts (pp. 195-210). New York, New York, USA: ACM Press.
- [Background] Pallavicini, F, Pepe, A., & Minissi, M. E. (2019). Gaming in Virtual Reality: What Changes in Terms of Usability, Emotional Response and Sense of Presence Compared to Non-Immersive Video Games? Simulation & Gaming, 104687811983142.
- [Background] Pallavicini F, Pepe A. Virtual Reality Games and the Role of Body Involvement in Enhancing Positive Emotions and Decreasing Anxiety: Within-Subjects Pilot Study. JMIR Serious Games. 2020 Jun 17;8(2):e15635. doi: 10.2196/15635. PMID 32554371
- [Background] Parong, J., Mayer, R. E., Fiorella, L., MacNamara, A., Homer, B. D., & Plass, J. L. (2017). Learning executive function skills by playing focused video games. Contemporary Educational Psychology, 51, 141-151.
- [Background] Pedram, S., Palmisano, S., Perez, P., Mursic, R., & Farrelly, M. (2020). Examining the potential of virtual reality to deliver remote rehabilitation. Computers in Human Behavior, 105, 106223.
- [Background] Pizzoli SFM, Mazzocco K, Triberti S, Monzani D, Alcaniz Raya ML, Pravettoni G. User-Centered Virtual Reality for Promoting Relaxation: An Innovative Approach. Front Psychol. 2019 Mar 12;10:479. doi: 10.3389/fpsyg.2019.00479. eCollection 2019. PMID 30914996
- [Background] Powers MB, Asmundson GJ, Smits JA. Exercise for Mood and Anxiety Disorders: The State-of-the Science. Cogn Behav Ther. 2015;44(4):237-9. doi: 10.1080/16506073.2015.1047286. No abstract available. PMID 26057087
- [Background] Qiu J, Shen B, Zhao M, Wang Z, Xie B, Xu Y. A nationwide survey of psychological distress among Chinese people in the COVID-19 epidemic: implications and policy recommendations. Gen Psychiatr. 2020 Mar 6;33(2):e100213. doi: 10.1136/gpsych-2020-100213. eCollection 2020. PMID 32215365
- [Background] Quesnel D, Riecke BE. Are You Awed Yet? How Virtual Reality Gives Us Awe and Goose Bumps. Front Psychol. 2018 Nov 9;9:2158. doi: 10.3389/fpsyg.2018.02158. eCollection 2018. PMID 30473673
- [Background] Repetto C, Gorini A, Vigna C, Algeri D, Pallavicini F, Riva G. The use of biofeedback in clinical virtual reality: the INTREPID project. J Vis Exp. 2009 Nov 12;(33):1554. doi: 10.3791/1554. PMID 19915521
- [Background] Riva G, Vigna C, Grassi A, Raspelli S, Cipresso P, Pallavicini F, Serino S, Gaggioli A. Learning Island: the development of a virtual reality system for the experiential training of stress management. Stud Health Technol Inform. 2012;173:369-71. PMID 22357020
- [Background] Riva G, Wiederhold BK. How Cyberpsychology and Virtual Reality Can Help Us to Overcome the Psychological Burden of Coronavirus. Cyberpsychol Behav Soc Netw. 2020 May;23(5):277-279. doi: 10.1089/cyber.2020.29183.gri. Epub 2020 Apr 17. No abstract available. PMID 32310689
- [Background] Rizzo A, Parsons TD, Lange B, Kenny P, Buckwalter JG, Rothbaum B, Difede J, Frazier J, Newman B, Williams J, Reger G. Virtual reality goes to war: a brief review of the future of military behavioral healthcare. J Clin Psychol Med Settings. 2011 Jun;18(2):176-87. doi: 10.1007/s10880-011-9247-2. PMID 21553133
- [Background] Rothbaum BO, Hodges LF, Kooper R, Opdyke D, Williford JS, North M. Effectiveness of computer-generated (virtual reality) graded exposure in the treatment of acrophobia. Am J Psychiatry. 1995 Apr;152(4):626-8. doi: 10.1176/ajp.152.4.626. PMID 7694917
- [Background] Shin M, Heard R, Suo C, Chow CM. Positive Emotions Associated with "Counter-Strike" Game Playing. Games Health J. 2012 Oct;1(5):342-7. doi: 10.1089/g4h.2012.0010. PMID 26192000
- [Background] Stetz MC, Kaloi-Chen JY, Turner DD, Bouchard S, Riva G, Wiederhold BK. The effectiveness of technology-enhanced relaxation techniques for military medical warriors. Mil Med. 2011 Sep;176(9):1065-70. doi: 10.7205/milmed-d-10-00393. PMID 21987967
- [Background] Valdez P, Mehrabian A. Effects of color on emotions. J Exp Psychol Gen. 1994 Dec;123(4):394-409. doi: 10.1037//0096-3445.123.4.394. PMID 7996122
- [Background] Walshe DG, Lewis EJ, Kim SI, O'Sullivan K, Wiederhold BK. Exploring the use of computer games and virtual reality in exposure therapy for fear of driving following a motor vehicle accident. Cyberpsychol Behav. 2003 Jun;6(3):329-34. doi: 10.1089/109493103322011641. PMID 12855091
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wechsler TF, Kumpers F, Muhlberger A. Inferiority or Even Superiority of Virtual Reality Exposure Therapy in Phobias?-A Systematic Review and Quantitative Meta-Analysis on Randomized Controlled Trials Specifically Comparing the Efficacy of Virtual Reality Exposure to Gold Standard in vivo Exposure in Agoraphobia, Specific Phobia, and Social Phobia. Front Psychol. 2019 Sep 10;10:1758. doi: 10.3389/fpsyg.2019.01758. eCollection 2019. PMID 31551840
- [Background] Zhu J, Sun L, Zhang L, Wang H, Fan A, Yang B, Li W, Xiao S. Prevalence and Influencing Factors of Anxiety and Depression Symptoms in the First-Line Medical Staff Fighting Against COVID-19 in Gansu. Front Psychiatry. 2020 Apr 29;11:386. doi: 10.3389/fpsyt.2020.00386. eCollection 2020. PMID 32411034
- [Derived] Pallavicini F, Orena E, Arnoldi L, Achille F, Stefanini S, Cassa M, Pepe A, Veronese G, Bernardelli L, Sforza F, Fascendini S, Defanti CA, Gemma M, Clerici M, Riva G, Mantovani F. Effects and Acceptability of a 1-Week Home-Based Virtual Reality Training for Supporting the Management of Stress and Anxiety: Randomized Pilot Trial. JMIR Serious Games. 2025 Mar 6;13:e50326. doi: 10.2196/50326. PMID 40053782
- [Derived] Pallavicini F, Orena E, di Santo S, Greci L, Caragnano C, Ranieri P, Vuolato C, Pepe A, Veronese G, Stefanini S, Achille F, Dakanalis A, Bernardelli L, Sforza F, Rossini A, Caltagirone C, Fascendini S, Clerici M, Riva G, Mantovani F. A virtual reality home-based training for the management of stress and anxiety among healthcare workers during the COVID-19 pandemic: study protocol for a randomized controlled trial. Trials. 2022 Jun 2;23(1):451. doi: 10.1186/s13063-022-06337-2. PMID 35655231
- See also: Johns Hopkins Coronavirus Resource Center. (2020). COVID-19 Map. — https://coronavirus.jhu.edu/map.html
- See also: World Health Organization. (2019). Occupational safety and health in public health emergencies: a manual for protecting health workers and responders. — https://www.who.int/publications/i/item/9789241514347